CLINICAL TRIAL: NCT02434042
Title: Study on Oral Administration of Bifidobacterium Longum BB536 on Incidence of Acute Diarrhea and/or Respiratory- Related Illnesses Compared to Placebo
Brief Title: Effects of Bifidobacterium Longum BB536 on Incidence of Acute Diarrhea and/or Respiratory- Related Illnesses in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Morinaga Milk Industry Co., LTD (Industry)
Responsible Party: Principal Investigator, Min-Tze LIONG, Associate Professor Dr, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 304/PTEKIND/650689
Record Dates: First submitted 2015-04-29; First posted 2015-05-05 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Healthy Volunteers
Keywords: probiotic; children; gastrointestinal; upper respiratory
MeSH Terms: interventions — Dextrins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BB536 (Active Comparator): Bifidobacterium longum BB536 (9 log CFU/day) and dextrin
  Interventions: Dietary Supplement: BB536
- Placebo (Placebo Comparator): 100% dextrin
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: BB536 — Intervention consists of daily administration of 1g probiotic Bifidobacterium longum BB536, administer daily for five days a week at a fixed dosage of 9 log CFU/day for BB536 and continue for 10 months.
  Other Names: Bifidobacterium longum BB536
  Arms: BB536
Other: Placebo — Intervention consists of daily administration of 1g of 100% dextrin, administer daily for five days a week and continue for 10 months.
  Other Names: 100% dextrin
  Arms: Placebo

SUMMARY:
This project aims to study the benefits of probiotics namely Bifidobacterium longum BB536 in prevention of acute diarrhea and/or respiratory-related illnesses, which are found common among children in Malaysia aged from 2 to 6 years.

DETAILED DESCRIPTION:
Data from WHO revealed that 5.2 million of children under five of age die every year due to preventable disease such as diarrhea, malaria and pneumonia. In Malaysia, reported cases of diarrhea and acute gastroenteritis have been observed to occur throughout the year, with rotavirus-associated diarrhea being the most prevalently identified gastrointestinal disorder.

Probiotics are preparations of bacteria and yeasts that are considered to confer a beneficial health effect when taken in an adequate amount. Bifidobacterium longum BB536, is a probiotic with over 100 scientific publications based on in vitro, in vivo, and clinical studies, with long consumption history supporting safety and health benefits.

BB536 is also commercially available in Malaysia and Japan in the form of food supplement and health supplements. Some of these include health supplements for children such as MAXBIOTICS, KidsBiotics and JANIPRO BB-G. All these three brands are sold in Malaysia and they all contain mixture of raw ingredient Bifidobacterium longum BB536 manufactured by Morinaga Milk Industry Co., Ltd. and other probiotic strains. In this study, the investigational product, Bifidobacterium longum BB536 and placebo is manufactured by Morinaga Milk Industry Co. Ltd., Japan.

Morinaga BB536 had been awarded FOSHU (Food for Specified Health Uses) status by Japan's Ministry of Health, Labour and Welfare. This status is granted to food products that have been shown in human clinical studies to demonstrate specific health benefits. Also, in year 2007, BB536 had obtained GRAS (Generally Recognised As Safe) certification in USA by FDA. BB536 has confirmed its safety for consumption as it is made in HACCP certified manufacturing plant (Pacific Resources, 2012). BB536 does not contain any porcine or bovine ingredients and has obtained the HALAL certification from the Japan Muslim Association (JMA), Japan. JMA is recognized by JAKIM, Malaysia.

Morinaga B. longum BB536 has been the subject of extensive clinical research and technical development with evidences from more than 100 scientific publications. There are no side effects been reported from the consumption of BB536 including premature infants, pregnant women, elderly people and patients who are taking immunosuppressive drugs. Based on in vitro, in vivo, and clinical studies, long consumption history (more than 30 years) support the safety and health benefits of the strain BB536 by improving intestinal environment, prevention of diarrhea, alleviation of constipation as well as supporting immune system. Based on previous study, ingestion of yogurt fortified with B. longum BB536 can help to reduce harmful bacteria such as Enterobacteriaceae, Streptococcus and C. perfringens, while at the same time alter the microbiota gut profile of volunteers with a significant increase of beneficial microbes Bifidobacterium and Lactobacillus species. Additionally, putrefactive substances in the intestinal environment were also reduced in the presence of the probiotic supplement. There was also clinical trial done on infants in Hidaka General Hospital through the administration of lyophilized powder containing B. longum BB536 and B. breve M-16V each at 9 log cfu/sachet. Such findings suggest that B. longum BB536 is safe and could be used further to evaluate its effect in preventing diarrhea and/or respiratory-related illness prevalence in children from daycare centres.

A total number of five hundred and twenty (520) healthy children from age 2-6 years old will be recruited for this study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male/ female subjects
* 2-6 years old
* BMI within a healthy range (between 5th to 84th percentile according to children BMI-for-age chart)
* Willing to commit throughout the experiment

Exclusion Criteria:

* Type-1 diabetes
* Long term medication due to certain severe illness
* HIV/AIDS
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 520 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2016-02-28 (Actual); Study Completion 2016-02-28 (Actual)

PRIMARY OUTCOMES:
Absentia between BB536 vs. Placebo children in daycare centers due to diarrhea and/or respiratory-related illnesses | 10 monhts
Severity of diarrhea between BB536 vs. Placebo children | 10 months
Severity of respiratory-related illnesses between BB536 vs. Placebo children | 10 months

SECONDARY OUTCOMES:
Fecal microbiota profiles of BB536 vs. Placebo children | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Min Tze Liong, PhD, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- School of Industrial Technology, Universiti Sains Malaysia, Pulau Pinang, Malaysia